CLINICAL TRIAL: NCT02377115
Title: Risk Assessment for Postoperative Delirium: Derivation of a Self-Administered Tablet Computer-based Clinical Screening Tool
Brief Title: Risk Assessment for Postoperative Delirium
Acronym: RAPID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Nicolai Goettel, Nicolai Goettel, MD, University Hospital, Basel, Switzerland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RAPID
Record Dates: First submitted 2015-02-14; First posted 2015-03-03 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Postoperative Delirium
Keywords: Postoperative delirium; Postoperative cognitive decline; Postoperative cognitive dysfunction; Risk assessment; Tablet computer; Clinical screening tool
MeSH Terms: conditions — Emergence Delirium; Postoperative Cognitive Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study cohort (Other): Tablet computer application
  Interventions: Other: Tablet computer application

INTERVENTIONS:
Other: Tablet computer application — Preoperatively, all study participants (entire cohort) will perform in the self-administered tablet computer-based tool to assess the risk of developing POD.

SUMMARY:
Postoperative delirium (POD) - a temporary state of confusion - is a frequent complication of surgery, which most commonly occurs in elderly patients. A tablet computer application that may assist preoperative risk screening for POD was developed at the University Hospital Basel in 2014. This study aims to investigate whether the computer program may assess the risk of a patient to develop POD.

DETAILED DESCRIPTION:
Background:

Postoperative delirium (POD) - a temporary state of confusion - is a frequent complication of surgery, which most commonly occurs in elderly patients. Depending on the risk profile, 9-87% of patients are affected. Regarding the increasing age of surgical patients, prevention of POD is of even greater importance. New data lead to the assumption that medical preventive strategies may influence the frequency or at least the severity or duration of POD.

Preventive measures in patients at increased risk for developing POD could possibly be administered; however, clinical predictors for POD are rare and/or unspecific. Different scores and test batteries to assess the preoperative risk of POD have been developed, but these tools are time-consuming and require trained personnel.

In 2014, a tablet computer application was developed at the University Hospital Basel with the primary objective to assess the risk of developing POD in surgical patients. The first part records patient details, such as age, level of training, language, sensory impairment, and regular drug intake. The second part tests different cognitive functions, more precisely cognitive self-assessment, temporal orientation, episodic memory, working memory, attention, and executive functions. In contrary to already available tools, this application can be operated by the patient alone without the help of trained staff. It was tested in healthy individuals and patients with mild cognitive impairment and should now be evaluated in a clinical setting.

Study design:

Prospective observational cohort study with a derivation cohort including patients scheduled for elective non-cardiac surgery.

Number of participants:

Patients will be enrolled until a collective of 50 patients with POD is reached. Each study participant in the collective of delirious patients represents 2% in the final analysis. With an expected incidence of POD of 25%, an overall sample size of about 200 patients will be recruited.

Recruitment:

Eligible study participants (patients scheduled for surgery at the University Hospital Basel) will be identified from the appointments calendar of the Anesthesia Preoperative Evaluation Clinic.

Methods:

Before surgery, participating patients perform the tablet computer application to obtain a score. A high score attained in the application suggests a low risk to develop POD. The score is then compared with results of postoperative assessments conducted daily from day 1 after surgery. Outcome measures are the Delirium-Rating-Scale-Revised-98 (DRS-R-98), which can be used to diagnose delirium and assess its severity, the Delirium Observation Screening (DOS) Scale, and the Confusion Assessment Method (CAM). These assessments are repeated for 5 days until the patient is discharged or - if the patient develops delirium - until symptoms have subsided.

Endpoints:

Primary endpoint:

Correlation between the test score attained by the patient in the self-administered computerized test and the incidence of POD.

Secondary endpoint:

Correlation between the test score attained by the patient in the self-administered computerized test and the severity of POD.

ELIGIBILITY:
Inclusion Criteria:

* Elective major surgery
* Age ≥65 years
* Education ≥7 years
* Fluency in German language
* Informed written consent

Exclusion Criteria:

* Dementia (Mini Mental State Examination (MMSE) <20 points)
* Surgical intervention that would limit verbal communication
* Cardiac surgery
* Thoracic/pulmonary surgery
* Intracranial surgery
* Former or present participation in a cognitive research project

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Incidence of POD. | Day 1-5 after surgery.
  Incidence of POD, detected by the DRS-R-98.

SECONDARY OUTCOMES:
Severity of POD. | Day 1-5 after surgery.
  Severity of POD, measured by the DRS-R-98.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolai Goettel, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schrader SL, Wellik KE, Demaerschalk BM, Caselli RJ, Woodruff BK, Wingerchuk DM. Adjunctive haloperidol prophylaxis reduces postoperative delirium severity and duration in at-risk elderly patients. Neurologist. 2008 Mar;14(2):134-7. doi: 10.1097/NRL.0b013e318166b88c. PMID 18332845
- [Background] Steiner LA. Postoperative delirium. Part 1: pathophysiology and risk factors. Eur J Anaesthesiol. 2011 Sep;28(9):628-36. doi: 10.1097/EJA.0b013e328349b7f5. PMID 21785356
- [Background] Dasgupta M, Hillier LM. Factors associated with prolonged delirium: a systematic review. Int Psychogeriatr. 2010 May;22(3):373-94. doi: 10.1017/S1041610209991517. Epub 2010 Jan 21. PMID 20092663
- [Background] Dasgupta M, Dumbrell AC. Preoperative risk assessment for delirium after noncardiac surgery: a systematic review. J Am Geriatr Soc. 2006 Oct;54(10):1578-89. doi: 10.1111/j.1532-5415.2006.00893.x. PMID 17038078
- [Background] Parente D, Luis C, Veiga D, Silva H, Abelha F. Congestive heart failure as a determinant of postoperative delirium. Rev Port Cardiol. 2013 Sep;32(9):665-71. doi: 10.1016/j.repc.2012.12.020. Epub 2013 Sep 6. PMID 24011864
- [Background] Zakriya KJ, Christmas C, Wenz JF Sr, Franckowiak S, Anderson R, Sieber FE. Preoperative factors associated with postoperative change in confusion assessment method score in hip fracture patients. Anesth Analg. 2002 Jun;94(6):1628-32, table of contents. doi: 10.1097/00000539-200206000-00050. PMID 12032042
- [Background] Kalisvaart KJ, Vreeswijk R, de Jonghe JF, van der Ploeg T, van Gool WA, Eikelenboom P. Risk factors and prediction of postoperative delirium in elderly hip-surgery patients: implementation and validation of a medical risk factor model. J Am Geriatr Soc. 2006 May;54(5):817-22. doi: 10.1111/j.1532-5415.2006.00704.x. PMID 16696749
- [Background] Marcantonio ER, Goldman L, Mangione CM, Ludwig LE, Muraca B, Haslauer CM, Donaldson MC, Whittemore AD, Sugarbaker DJ, Poss R, et al. A clinical prediction rule for delirium after elective noncardiac surgery. JAMA. 1994 Jan 12;271(2):134-9. PMID 8264068
- [Background] Inouye SK, Viscoli CM, Horwitz RI, Hurst LD, Tinetti ME. A predictive model for delirium in hospitalized elderly medical patients based on admission characteristics. Ann Intern Med. 1993 Sep 15;119(6):474-81. doi: 10.7326/0003-4819-119-6-199309150-00005. PMID 8357112
- [Background] Freter SH, Dunbar MJ, MacLeod H, Morrison M, MacKnight C, Rockwood K. Predicting post-operative delirium in elective orthopaedic patients: the Delirium Elderly At-Risk (DEAR) instrument. Age Ageing. 2005 Mar;34(2):169-71. doi: 10.1093/ageing/afh245. No abstract available. PMID 15713861
- [Background] Rudolph JL, Jones RN, Levkoff SE, Rockett C, Inouye SK, Sellke FW, Khuri SF, Lipsitz LA, Ramlawi B, Levitsky S, Marcantonio ER. Derivation and validation of a preoperative prediction rule for delirium after cardiac surgery. Circulation. 2009 Jan 20;119(2):229-36. doi: 10.1161/CIRCULATIONAHA.108.795260. Epub 2008 Dec 31. PMID 19118253
- [Background] Long LS, Shapiro WA, Leung JM. A brief review of practical preoperative cognitive screening tools. Can J Anaesth. 2012 Aug;59(8):798-804. doi: 10.1007/s12630-012-9737-1. Epub 2012 May 26. PMID 22638676
- [Background] Egerhazi A, Berecz R, Bartok E, Degrell I. Automated Neuropsychological Test Battery (CANTAB) in mild cognitive impairment and in Alzheimer's disease. Prog Neuropsychopharmacol Biol Psychiatry. 2007 Apr 13;31(3):746-51. doi: 10.1016/j.pnpbp.2007.01.011. Epub 2007 Jan 16. PMID 17289240
- [Background] Erlanger DM, Kaushik T, Broshek D, Freeman J, Feldman D, Festa J. Development and validation of a web-based screening tool for monitoring cognitive status. J Head Trauma Rehabil. 2002 Oct;17(5):458-76. doi: 10.1097/00001199-200210000-00007. PMID 12802255
- [Background] Fillit HM, Simon ES, Doniger GM, Cummings JL. Practicality of a computerized system for cognitive assessment in the elderly. Alzheimers Dement. 2008 Jan;4(1):14-21. doi: 10.1016/j.jalz.2007.09.008. PMID 18631946
- [Background] Levinson D, Reeves D, Watson J, Harrison M. Automated neuropsychological assessment metrics (ANAM) measures of cognitive effects of Alzheimer's disease. Arch Clin Neuropsychol. 2005 May;20(3):403-8. doi: 10.1016/j.acn.2004.09.001. PMID 15797175
- [Background] Saxton J, Morrow L, Eschman A, Archer G, Luther J, Zuccolotto A. Computer assessment of mild cognitive impairment. Postgrad Med. 2009 Mar;121(2):177-85. doi: 10.3810/pgm.2009.03.1990. PMID 19332976
- [Background] Falleti MG, Maruff P, Collie A, Darby DG. Practice effects associated with the repeated assessment of cognitive function using the CogState battery at 10-minute, one week and one month test-retest intervals. J Clin Exp Neuropsychol. 2006 Oct;28(7):1095-112. doi: 10.1080/13803390500205718. PMID 16840238
- [Background] Tornatore JB, Hill E, Laboff JA, McGann ME. Self-administered screening for mild cognitive impairment: initial validation of a computerized test battery. J Neuropsychiatry Clin Neurosci. 2005 Winter;17(1):98-105. doi: 10.1176/jnp.17.1.98. PMID 15746489
- [Background] Wild K, Howieson D, Webbe F, Seelye A, Kaye J. Status of computerized cognitive testing in aging: a systematic review. Alzheimers Dement. 2008 Nov;4(6):428-37. doi: 10.1016/j.jalz.2008.07.003. PMID 19012868
- [Background] Elwood RW. MicroCog: assessment of cognitive functioning. Neuropsychol Rev. 2001 Jun;11(2):89-100. doi: 10.1023/a:1016671201211. PMID 11572473
- [Background] Gualtieri CT, Johnson LG. Reliability and validity of a computerized neurocognitive test battery, CNS Vital Signs. Arch Clin Neuropsychol. 2006 Oct;21(7):623-43. doi: 10.1016/j.acn.2006.05.007. Epub 2006 Oct 2. PMID 17014981
- [Background] Iverson GL, Brooks BL, Ashton VL, Johnson LG, Gualtieri CT. Does familiarity with computers affect computerized neuropsychological test performance? J Clin Exp Neuropsychol. 2009 Jul;31(5):594-604. doi: 10.1080/13803390802372125. Epub 2008 Oct 29. PMID 18972312
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Trzepacz PT, Mittal D, Torres R, Kanary K, Norton J, Jimerson N. Validation of the Delirium Rating Scale-revised-98: comparison with the delirium rating scale and the cognitive test for delirium. J Neuropsychiatry Clin Neurosci. 2001 Spring;13(2):229-42. doi: 10.1176/jnp.13.2.229. PMID 11449030
- [Background] Fratiglioni L, Jorm AF, Grut M, Viitanen M, Holmen K, Ahlbom A, Winblad B. Predicting dementia from the Mini-Mental State Examination in an elderly population: the role of education. J Clin Epidemiol. 1993 Mar;46(3):281-7. doi: 10.1016/0895-4356(93)90076-d. PMID 8455053
- [Background] Adamis D, Rooney S, Meagher D, Mulligan O, McCarthy G. A comparison of delirium diagnosis in elderly medical inpatients using the CAM, DRS-R98, DSM-IV and DSM-5 criteria. Int Psychogeriatr. 2015 Jun;27(6):883-9. doi: 10.1017/S1041610214002853. Epub 2015 Jan 20. PMID 25601222
- [Background] Grover S, Kate N. Assessment scales for delirium: A review. World J Psychiatry. 2012 Aug 22;2(4):58-70. doi: 10.5498/wjp.v2.i4.58. PMID 24175169
- [Background] Carvalho JP, de Almeida AR, Gusmao-Flores D. Delirium rating scales in critically ill patients: a systematic literature review. Rev Bras Ter Intensiva. 2013 Apr-Jun;25(2):148-54. doi: 10.5935/0103-507X.20130026. PMID 23917980
- [Background] Koster S, Hensens AG, Oosterveld FG, Wijma A, van der Palen J. The delirium observation screening scale recognizes delirium early after cardiac surgery. Eur J Cardiovasc Nurs. 2009 Oct;8(4):309-14. doi: 10.1016/j.ejcnurse.2009.02.006. Epub 2009 Mar 12. PMID 19285452
- See also: Delirium: diagnosis, prevention and management — http://www.guideline.gov/content.aspx?id=24121